CLINICAL TRIAL: NCT01890031
Title: The Interactive Cholesterol Advisory Tool
Brief Title: Interactive Cholesterol Advisory Tool
Acronym: ICAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Robert Block, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1R44HL097506-01 (NIH)
Record Dates: First submitted 2012-06-18; First posted 2013-07-01 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-08

CONDITIONS: Low Risk (0-10% Chance) of Developing Cardiovascular Disease Within 10 Years Based on Risk Factors; Moderate Risk (10-20% Chance) of Developing Cardiovascular (Heart) Disease Within 10 Years Based on Risk Factors
Keywords: cardiovascular disease; cholesterol
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Low Risk, No ICAT (No Intervention): Low risk, not randomized to use the Interactive Cholesterol Advisory Tool, no study physician visits
- Low risk, ICAT (Other): Low risk, randomized to use the Interactive Cholesterol Advisory Tool, no study physician visits
  Interventions: Other: Interactive Cholesterol Advisory Tool
- Low risk, ICAT, and study physician (Other): Low risk, assigned to use the Interactive Cholesterol Advisory Tool, and study physician visits.
  Interventions: Other: Interactive Cholesterol Advisory Tool; Other: Study physician visits
- Moderate risk, no ICAT (Other): Moderate risk, study physician visits, and not randomized to use the Interactive Cholesterol Advisory Tool
  Interventions: Other: Study physician visits
- Moderate risk, ICAT (Other): Moderate risk, study physician visits, and randomized to use the Interactive Cholesterol Advisory Tool
  Interventions: Other: Interactive Cholesterol Advisory Tool; Other: Study physician visits

INTERVENTIONS:
Other: Interactive Cholesterol Advisory Tool — using the virtual clinician computer program for cholesterol information and education.
  Arms: Low risk, ICAT; Low risk, ICAT, and study physician; Moderate risk, ICAT
Other: Study physician visits — In-person individual visits with a study physician to give information on cholesterol
  Arms: Low risk, ICAT, and study physician; Moderate risk, ICAT; Moderate risk, no ICAT

SUMMARY:
The purpose of this study is to show that we can effectively deliver health information and education, online, via computer regarding cholesterol. This computer program is called the Interactive Cholesterol Advisory Tool (ICAT).

DETAILED DESCRIPTION:
Participants will be recruited and categorized based on screening labs into 1 of 2 groups: Low or moderate risk of developing cardiovascular disease within 10 years based on risk factors. The low risk group will be advised to take the blood test results furnished by the study to their primary care doctor to discuss managing cholesterol. The moderate risk group will see the study physician for 4 visits about high cholesterol. Both groups complete a total of 4 blood draws over 9 months. Both groups will be randomized at consent into 2 groups: 1 who uses the Interactive Cholesterol Advisory Tool (ICAT) and 1 that does not use the ICAT. Because recruitment goals for the low risk group were met, a third group was created: low risk who both the study physician for 4 visits about high cholesterol and use the ICAT.

ELIGIBILITY:
Inclusion Criteria:

* Fluency in English,
* Willing to come in for 1-5 visits,
* Low and moderate CVD risk.
* Having access to a computer with internet connection

Exclusion Criteria:

* CVD diagnosis or CVD equivalent,
* Psychosis, terminal illness,
* Pregnancy,
* Current statin use if assigned to the low risk group
* Liver disease,
* Peripheral Vascular Disease,
* Diabetes Mellitus,
* Abdominal Aortic Aneurism,
* Cerebral Vascular Disease
* Triglyceride level above 500 mg/dl
* Uncorrected hypothyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Block, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Block RC, Abdolahi A, Niemiec CP, Rigby CS, Williams GC. Effects of an evidence-based computerized virtual clinician on low-density lipoprotein and non-high-density lipoprotein cholesterol in adults without cardiovascular disease: The Interactive Cholesterol Advisory Tool. Health Informatics J. 2016 Dec;22(4):897-910. doi: 10.1177/1460458215600040. Epub 2015 Aug 21. PMID 26297222

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Risk, No ICAT | Low Risk, ICAT | Moderate Risk, no ICAT | Moderate Risk, ICAT | Low Risk, ICAT, and Study Physician
Started | 50 | 50 | 12 | 11 | 8
Completed | 50 | 50 | 12 | 11 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk, No ICAT | Low Risk, ICAT | Moderate Risk, no ICAT | Moderate Risk, ICAT | Low Risk, ICAT, and Study Physician | Total
Number analyzed (Participants) | 50 | 50 | 12 | 11 | 8 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11.9) | 46.6 (13.5) | 53.3 (9.7) | 57.7 (8.8) | 51.4 (13.0) | 49.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 5 | 3 | 7 | 86
  Male | 12 | 17 | 7 | 8 | 1 | 45
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 12 | 11 | 8 | 131
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 125.5 (31.4) | 123.3 (32.5) | 130.4 (37.8) | 121.2 (41.7) | 129.9 (38.2) | 125.7 (33.4)

OUTCOME MEASURES:

1. Primary Outcome: LDL-C in All ICAT Group Participants Versus Non-ICAT Group Participants
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Risk, No ICAT | Low Risk, ICAT | Moderate Risk, no ICAT | Moderate Risk, ICAT | Low Risk, ICAT, and Study Physician
Number analyzed (Participants) | 50 | 50 | 12 | 11 | 8
mg/dL | 126.2 (32.3) | 126.0 (28.8) | 103.2 (35.1) | 107.7 (32.3) | 107.0 (45.7)

2. Secondary Outcome: Number of Participants Who Adhered to Medication Prescribed as Self Reported at 9 Months
Description: We will assess adherence (for those who are prescribed a statin in the moderate CVD risk group) by both indirect objective measures and subjective reports. The study design did not include prescription of a cholesterol-lowering medication as per randomization. Participants were prescribed a statin as standard of care based on the participants and physicians agreement. Low risk individuals have less need for medication compared to moderate risk based on the current science.
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | Low Risk, No ICAT | Low Risk, ICAT | Moderate Risk, no ICAT | Moderate Risk, ICAT | Low Risk, ICAT, and Study Physician
Number analyzed (Participants) | 50 | 50 | 12 | 11 | 8
participants | 2 | 1 | 9 | 7 | 0

ADVERSE EVENTS:
Time Frame: Data were collected at over 9 months.
Arm/Group | Low Risk, No ICAT | Low Risk, ICAT | Moderate Risk, no ICAT | Moderate Risk, ICAT | Low Risk, ICAT, and Study Physician
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/12 | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/12 | 0/11 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No